CLINICAL TRIAL: NCT03369574
Title: Prospective Observational Study of Chronic Rhinosinusitis Symptoms in Asthma Patients Undergoing Treatment With Reslizumab
Brief Title: Study of Chronic Rhinosinusitis Symptoms in Asthma Patients Undergoing Treatment With Reslizumab
Status: Withdrawn | Type: Observational
Why Stopped: Study personnel diverted to other activities and the study was not commenced
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Li-Xing Man, Associate Professor, University of Rochester
Other Study IDs: RSRB 60712
Record Dates: First submitted 2017-12-02; First posted 2017-12-12 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Chronic Rhinosinusitis (Diagnosis); Asthma; Nasal Polyps
MeSH Terms: conditions — Disease; Asthma; Nasal Polyps | interventions — reslizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- chronic rhinosinusitis and eosinophilic asthma: Adults over the age of 18, diagnosed with poorly controlled moderate to severe asthma with an eosinophilic phenotype (defined by blood eosinophil count of 150 µL or greater within 6 weeks of enrollment) who are initiating/undergoing reslizumab therapy and also carry a physician diagnosis of chronic rhinosinusitis with nasal polyposis
  Interventions: Drug: Reslizumab

INTERVENTIONS:
Drug: Reslizumab — reslizumab administration

SUMMARY:
The primary objective of this research is to monitor chronic rhinosinusitis (CRS) symptoms in asthma patients who are undergoing treatment with reslizumab. A secondary objective is to explore whether there are sub-populations that appear to benefit or not benefit from reslizumab in terms of their CRS symptoms.

DETAILED DESCRIPTION:
This is a prospective observational study of patients receiving reslizumab to treat their asthma. Some asthma patients receiving reslizumab also have CRS, which might also be improved by this drug. Study measures will be obtained from the medical records of eligible subjects who consent to participate. The study has no specific procedures per se, because all study measures are acquired during the course of standard of care treatment and will be abstracted from those medical records.

ELIGIBILITY:
Inclusion Criteria:

* Age is 18 years or older
* Physician diagnosis of poorly controlled moderate to severe asthma despite typical medical therapy with an eosinophilic phenotype (defined by blood eosinophil count of 150 µL or greater within 6 weeks of enrollment)
* Initiating or undergoing reslizumab therapy (Reslizumab - Patient Information listed in Appendix 1 for reference)
* Physician diagnosis of chronic rhinosinusitis with nasal polyposis
* Able to understand and willing to provide informed consent
* Able to complete standard of care English-language questionnaires

Exclusion Criteria:

* Current smokers
* Significant uncontrolled medical conditions
* Ongoing malignancy or history of cancer in remission for less than 12 months
* Subjects who had received immunosuppressive medications within 3 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with poorly controlled moderate to severe asthma with eosinophilia and a diagnosis of chronic rhinosinusitis with nasal polyposis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Mean Sino-Nasal Outcome Test (SNOT)-22 Score | 1 year
  SNOT-22 score ranges from 0 to 110 with higher scores indicating worse symptoms. The questionnaire consists of 22 questions regarding common sinonasal complaints of patients with chronic sinus disease, each question graded 0 to 5 (0 No Problem, 1 Very Mild Problem, 2 Mild or Slight Problem, 3 Moderate Problem, 4 Severe Problem, 5 Problem as Bad as it Can Be).

CONTACTS AND LOCATIONS:
Overall Officials: Li-Xing Man, MSc, MD, MPA, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Department of Otolaryngology Head and Neck Surgery, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hastan D, Fokkens WJ, Bachert C, Newson RB, Bislimovska J, Bockelbrink A, Bousquet PJ, Brozek G, Bruno A, Dahlen SE, Forsberg B, Gunnbjornsdottir M, Kasper L, Kramer U, Kowalski ML, Lange B, Lundback B, Salagean E, Todo-Bom A, Tomassen P, Toskala E, van Drunen CM, Bousquet J, Zuberbier T, Jarvis D, Burney P. Chronic rhinosinusitis in Europe--an underestimated disease. A GA(2)LEN study. Allergy. 2011 Sep;66(9):1216-23. doi: 10.1111/j.1398-9995.2011.02646.x. Epub 2011 May 24. PMID 21605125
- [Background] Hamilos DL. Chronic rhinosinusitis: epidemiology and medical management. J Allergy Clin Immunol. 2011 Oct;128(4):693-707; quiz 708-9. doi: 10.1016/j.jaci.2011.08.004. Epub 2011 Sep 3. PMID 21890184
- [Background] Rosenfeld RM, Piccirillo JF, Chandrasekhar SS, Brook I, Ashok Kumar K, Kramper M, Orlandi RR, Palmer JN, Patel ZM, Peters A, Walsh SA, Corrigan MD. Clinical practice guideline (update): adult sinusitis. Otolaryngol Head Neck Surg. 2015 Apr;152(2 Suppl):S1-S39. doi: 10.1177/0194599815572097. PMID 25832968
- [Background] Settipane GA, Chafee FH. Nasal polyps in asthma and rhinitis. A review of 6,037 patients. J Allergy Clin Immunol. 1977 Jan;59(1):17-21. doi: 10.1016/0091-6749(77)90171-3. PMID 833373
- [Background] Jarvis D, Newson R, Lotvall J, Hastan D, Tomassen P, Keil T, Gjomarkaj M, Forsberg B, Gunnbjornsdottir M, Minov J, Brozek G, Dahlen SE, Toskala E, Kowalski ML, Olze H, Howarth P, Kramer U, Baelum J, Loureiro C, Kasper L, Bousquet PJ, Bousquet J, Bachert C, Fokkens W, Burney P. Asthma in adults and its association with chronic rhinosinusitis: the GA2LEN survey in Europe. Allergy. 2012 Jan;67(1):91-8. doi: 10.1111/j.1398-9995.2011.02709.x. Epub 2011 Nov 4. PMID 22050239
- [Background] Bachert C, Zhang N, Holtappels G, De Lobel L, van Cauwenberge P, Liu S, Lin P, Bousquet J, Van Steen K. Presence of IL-5 protein and IgE antibodies to staphylococcal enterotoxins in nasal polyps is associated with comorbid asthma. J Allergy Clin Immunol. 2010 Nov;126(5):962-8, 968.e1-6. doi: 10.1016/j.jaci.2010.07.007. PMID 20810157
- [Background] Bachert C, Gevaert P, Holtappels G, Cuvelier C, van Cauwenberge P. Nasal polyposis: from cytokines to growth. Am J Rhinol. 2000 Sep-Oct;14(5):279-90. doi: 10.2500/105065800781329573. PMID 11068652
- [Background] Bachert C, Wagenmann M, Hauser U, Rudack C. IL-5 synthesis is upregulated in human nasal polyp tissue. J Allergy Clin Immunol. 1997 Jun;99(6 Pt 1):837-42. doi: 10.1016/s0091-6749(97)80019-x. PMID 9215253
- [Background] Bousquet J, Chanez P, Lacoste JY, Barneon G, Ghavanian N, Enander I, Venge P, Ahlstedt S, Simony-Lafontaine J, Godard P, et al. Eosinophilic inflammation in asthma. N Engl J Med. 1990 Oct 11;323(15):1033-9. doi: 10.1056/NEJM199010113231505. PMID 2215562
- [Background] Sanderson CJ. Interleukin-5, eosinophils, and disease. Blood. 1992 Jun 15;79(12):3101-9. No abstract available. PMID 1596561
- [Background] Takatsu K, Nakajima H. IL-5 and eosinophilia. Curr Opin Immunol. 2008 Jun;20(3):288-94. doi: 10.1016/j.coi.2008.04.001. Epub 2008 May 27. PMID 18511250
- [Background] Leckie MJ, ten Brinke A, Khan J, Diamant Z, O'Connor BJ, Walls CM, Mathur AK, Cowley HC, Chung KF, Djukanovic R, Hansel TT, Holgate ST, Sterk PJ, Barnes PJ. Effects of an interleukin-5 blocking monoclonal antibody on eosinophils, airway hyper-responsiveness, and the late asthmatic response. Lancet. 2000 Dec 23-30;356(9248):2144-8. doi: 10.1016/s0140-6736(00)03496-6. PMID 11191542
- [Background] Kips JC, O'Connor BJ, Langley SJ, Woodcock A, Kerstjens HA, Postma DS, Danzig M, Cuss F, Pauwels RA. Effect of SCH55700, a humanized anti-human interleukin-5 antibody, in severe persistent asthma: a pilot study. Am J Respir Crit Care Med. 2003 Jun 15;167(12):1655-9. doi: 10.1164/rccm.200206-525OC. Epub 2003 Mar 20. PMID 12649124
- [Background] Green RH, Brightling CE, McKenna S, Hargadon B, Parker D, Bradding P, Wardlaw AJ, Pavord ID. Asthma exacerbations and sputum eosinophil counts: a randomised controlled trial. Lancet. 2002 Nov 30;360(9347):1715-21. doi: 10.1016/S0140-6736(02)11679-5. PMID 12480423
- [Background] Jayaram L, Pizzichini MM, Cook RJ, Boulet LP, Lemiere C, Pizzichini E, Cartier A, Hussack P, Goldsmith CH, Laviolette M, Parameswaran K, Hargreave FE. Determining asthma treatment by monitoring sputum cell counts: effect on exacerbations. Eur Respir J. 2006 Mar;27(3):483-94. doi: 10.1183/09031936.06.00137704. PMID 16507847
- [Background] Nair P, Pizzichini MM, Kjarsgaard M, Inman MD, Efthimiadis A, Pizzichini E, Hargreave FE, O'Byrne PM. Mepolizumab for prednisone-dependent asthma with sputum eosinophilia. N Engl J Med. 2009 Mar 5;360(10):985-93. doi: 10.1056/NEJMoa0805435. PMID 19264687
- [Background] Castro M, Mathur S, Hargreave F, Boulet LP, Xie F, Young J, Wilkins HJ, Henkel T, Nair P; Res-5-0010 Study Group. Reslizumab for poorly controlled, eosinophilic asthma: a randomized, placebo-controlled study. Am J Respir Crit Care Med. 2011 Nov 15;184(10):1125-32. doi: 10.1164/rccm.201103-0396OC. Epub 2011 Aug 18. PMID 21852542
- [Background] Gevaert P, Bachert C, Holtappels G, Novo CP, Van der Heyden J, Fransen L, Depraetere S, Walter H, van Cauwenberge P, Tavernier J. Enhanced soluble interleukin-5 receptor alpha expression in nasal polyposis. Allergy. 2003 May;58(5):371-9. doi: 10.1034/j.1398-9995.2003.00110.x. PMID 12752323
- [Background] Simon HU, Yousefi S, Schranz C, Schapowal A, Bachert C, Blaser K. Direct demonstration of delayed eosinophil apoptosis as a mechanism causing tissue eosinophilia. J Immunol. 1997 Apr 15;158(8):3902-8. PMID 9103460